CLINICAL TRIAL: NCT01389518
Title: Evaluation of the Efficacy and Safety of Fixed Combination of Paracetamol, Chlorpheniramine and Phenylephrine in the Treatment of Symptomatic Common Cold and Flu Syndrome in Adults
Brief Title: Efficacy and Safety of Paracetamol, Chlorpheniramine and Phenylephrine in the Treatment of Common Cold and Flu Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Paulo Dornelles Picon, Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 05-492
Record Dates: First submitted 2011-02-15; First posted 2011-07-08 (Estimated); Last update posted 2011-11-28 (Estimated); Status verified 2011-11

CONDITIONS: Flu
Keywords: Symptomatic treatment; Common Cold; flu syndrome
MeSH Terms: conditions — Influenza, Human; Common Cold | interventions — Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Paracetamol,Chlorpheniramin,Phenylephrin (Active Comparator)
  Interventions: Drug: Active
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Active — 1 capsule de active (fixed combination of acetaminophen, chlorpheniramine and phenylephrine) administered in four 4-hour period of wakefulness in between at 07:00 and 23:00 (five daily doses) for two or three consecutive days
  Other Names: Active Flu
  Arms: Paracetamol,Chlorpheniramin,Phenylephrin
Drug: Placebo — 1 capsule administered in four 4-hour period of wakefulness in between at 07:00 and 23:00 (five daily doses) for two or three consecutive days
  Other Names: Placebo Comparator Flu
  Arms: Placebo

SUMMARY:
The aim of this study is to evaluate the efficacy and safety of a fixed combination of paracetamol, phenylephrine and chlorpheniramine in symptomatic treatment of common cold and flu-like illness in adults in a randomized, double-blind, controlled trial. The investigators included 146 healthy study subjects aged between 18 and 60 years who presented flu or common cold moderate to severe onset of less than 3 days (72 hours). After clinical and laboratory evaluation were randomized to receive active drug or placebo, five capsules a day, every 4 hours for 48-72h.The outcomes to assess the effectiveness involve the measurement of symptom scores, overall duration of symptoms, return to usual activities, use of rescue medication, improvement of the fever.

DETAILED DESCRIPTION:
The upper respiratory infections are frequent in the population, and its treatment, in most cases involves the use of symptomatic drugs. Paracetamol is used as an analgesic and antipyretic, whereas chlorpheniramine and phenylephrine is an antihistamine with a vasoconstrictor decongestant function. The aim of this study is to evaluate the efficacy and safety of a fixed combination of paracetamol, phenylephrine and chlorpheniramine in symptomatic treatment of common cold and flu-like illness in adults in a randomized, double-blind, controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* Men and women between 18 and 60;
* Presented symptoms of recent onset, for more than 6 hours and less than 72 hours, characterizing one of the following conditions:

the common cold, which consists of at least 2 symptoms among the 10 following: sneezing, rhinorrhea, nasal congestion, headache, muscle pain, discomfort in the throat, sore throat, dysphonia, cough, fever, the latter being of moderate to severe intensity through a symptom severity scale of 4 points (0 = none, 1 = mild, 2 = moderate, 3 = severe).

the flu syndrome, which consists of fever of at least 38.1 ° C and headache of moderate or severe intensity or myalgia / arthralgia moderate or severe using a scale of severity of symptoms of 4 points (0 = none, 1 = mild, 2 = moderate, 3 = severe).

* Adequate contraception if women of childbearing age.
* Ability to not use any other drugs for the treatment of clinical symptoms, except in cases of urgency, and immediate communication with the investigator, patients with chronic diseases being treated with monotherapy, stable over the past three months, could be included.
* Good understanding capacity and collaboration.
* Compliance with the informed consent form had been signed.

Exclusion Criteria:

* Pregnant women or nursing mothers
* Known hypersensitivity to components of the formula of anti-flu drug
* Use of alcohol or illicit drug use
* Use of monoamine oxidase inhibitors or barbiturates
* Diagnosis of seasonal or perennial allergic rhinitis in activity
* Presenting the diagnosis of any disease activity in acute or chronic disease exacerbated (uncompensated), including hypertension, ischemic heart disease, narrow-angle glaucoma, symptomatic prostatic hyperplasia, chronic renal failure, liver diseases, infectious tracheobronchitis presumably bacterial pneumonia, pharyngitis strep, asthma or chronic obstructive pulmonary disease and any disease or condition that in the opinion of the investigator can modify the results of their study is not due to the drug under investigation or that puts the patient at significant risk;
* Clinical evidence of immunosuppression;
* Patients who received influenza vaccine for the week prior to inclusion
* Patients who in the opinion of the attending physician and / or the investigator may need to receive antiviral drugs for treatment of infection with influenza virus A or B (eg, amantadine, rimantadine, oseltamivir, zanamivir)
* Patients who in the opinion of the attending physician and / or the investigator need receive antibacterial drugs for the treatment of acute respiratory infection
* Use of drugs prior to inclusion by time intervals of less than two doses of these drugs (in the case of associations, considered as the reference half-life longer): analgesics, nonsteroidal anti-inflammatory drugs, glucocorticoids and other immunosuppressants, antihistamines, Topical and systemic decongestants, and any medication that in the opinion of the investigator can modify the results of their study is not due to the drug under investigation or by an interaction that place the patient at significant risk
* Participation in another clinical research for less than a year.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 146 (Actual)
Dates: Start 2009-05; Primary Completion 2009-07 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Symptom score | 72 hours
  We assessed symptoms of common cold or flu-like illness with symptoms of global scale for assessing efficacy in clinical trial. The scale consists of 10 symptoms (sneezing, rhinorrhea, nasal congestion, headache, muscle pain, discomfort in the throat, sore throat, dysphonia, cough and fever). We used a Likert scale of intensity of 4 points where 0 no symptoms, 1 mild symptom, 2 moderate symptom, 3 severe symptom intensity.Overall duration of symptoms. Return to normal activity. Use of rescue medication for relief of symptoms. Improves fever by reducing the axillary temperature below 38.1 ° C

SECONDARY OUTCOMES:
Adverse events | 72 hours
  The safety of the product will be accompanied by subjective report of patients, the emergence of adverse effects such as drowsiness, nausea, eye pain, dizziness and palpitations. In addition, there will be accompanied by clinical laboratory parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Paulo D Piccon, Prof. Dr., Principal Investigator — Federal University of Rio Grande do Sul (UFRGS) / Hospital de Clinicas de Porto Alegre; Marisa B Costa, MS, Study Director — Federal University of Rio Grande do Sul; Luis Felipe C Schmidt, MD, Study Director — Hospital de Clinicas de Porto Alegre

REFERENCES:
- [Derived] Picon PD, Costa MB, da Veiga Picon R, Fendt LC, Suksteris ML, Saccilotto IC, Dornelles AD, Schmidt LF. Symptomatic treatment of the common cold with a fixed-dose combination of paracetamol, chlorphenamine and phenylephrine: a randomized, placebo-controlled trial. BMC Infect Dis. 2013 Nov 22;13:556. doi: 10.1186/1471-2334-13-556. PMID 24261438